CLINICAL TRIAL: NCT05711420
Title: Comparison of the Effects of the Education Given to Nursing Students by Gamification Method and Flipped Learning Method on the Level of Participation, Attitude, Interest and Motivation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sakarya University (Other)
Responsible Party: Principal Investigator, Metin Yildiz, Nurse (Asst.Prof.Dr.), Sakarya University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SakaryaU-metinyildiz-002
Record Dates: First submitted 2023-01-16; First posted 2023-02-03 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Educational Problems
Keywords: Gamification; Flipped learning; Interest; Motivation; Participation; Attitude
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Gamification method group (Experimental): The group to be trained by gamification method; A gamification application was made every week. Points are given in the table prepared for those who are successful in weekly participation in gamification, coming to the lesson with their homework done, participating in the discussions in the lesson, and in the evaluation at the end of the lesson. Every week, the winner was given a gift. At the end of the lesson, the points in the headings of "Leaderboard", "Badge" and "Status", which are the elements of the gamification method, were added weekly. And in the last week, a meeting was held with the students according to all scores and a post-test was applied.
  Interventions: Behavioral: Gamification method group
- Flipped learning group (Experimental): Before the study, videos were found each week that lecture on the relevant subject, videos were shot on the subject, and the videos were transferred to the students via a platform. At the end of each video, they were told to complete the homework on the subject and come to the lesson.
  In the lesson, the lesson was processed with activities according to the videos.
  Interventions: Behavioral: Flipped learning group
- Control group (No Intervention): Lessons were taught with traditional learning method.

INTERVENTIONS:
Behavioral: Gamification method group — Gamification method group
  Arms: Gamification method group
Behavioral: Flipped learning group — Flipped learning group
  Arms: Flipped learning group

SUMMARY:
In this study, it is aimed to compare the effects of the education given to nursing students with the gamification method and the flipped learning method on the level of participation, attitude, interest and motivation.

The research was conducted as a randomized controlled experimental study. The study population consisted of 110 student between October 2022 and January 2023, and the sample of the research consisted of 90 individuals selected from the population using the improbable random sampling method. "Descriptive Feature Form," "Teaching Material Motivation Scale," "Course Interest Scale", Attitude Scale Towards Learning and ''absence charts'' were used to collect data.

In the analysis of data; percentile distribution, chi-square, Fisher- Exact test, t-test in independent groups, Repeated Measures ANOVA Test, One Way ANOVA test, and post hoc analyzes (Bonferroni, Games Howell) were used.

ELIGIBILITY:
Inclusion Criteria:

* To be a student,
* 18 years and older
* Volunteer

Exclusion Criteria:

* Students who are not required to attend the course are not included.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2022-10-18 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-01-15 (Actual)

PRIMARY OUTCOMES:
Teaching Material Motivation Scale | Evaluated at the end of 6 weeks
  Teaching Material Motivation Instructional Material Motivation Scale: It was developed to measure the effect of instructional materials on students' motivation. The scale is a 5-point Likert-type scale consisting of 36 items. Each item in the scale will be scored from 1 (Not True) to 5 (Very True) by the students. Accordingly, the lowest score on the scale is 36, and the highest score is 180.
  In the Turkish adaptation study conducted by Acar (2009), the reliability coefficient (Cronbach Alpha value) was found to be 0.92 in the reliability analysis of the scale. An increase in the score on the scale indicates an increase in motivation.
Student Interest Scale | Evaluated at the end of 6 weeks
  Student Interest Scale; Developed by (Mazer, 2013) in order to evaluate its relationship with variables such as learning motivation, effective learning, and level of participation in the lesson, the Class Interest Scale is a 5-point Likert-type measurement tool consisting of 16 items and two sub-dimensions (affective and cognitive interest). et al (2015) ("1" Strongly disagree, "2" Disagree, "3" Undecided, "4" Agree, "5" Totally Agree). There is no reverse coded item in the scale. Affective interest sub-dimension of the scale consists of 9 items and cognitive interest sub-dimension consists of 7 items. The Cronbach's alpha internal consistency reliability coefficients of the scale were .95 for affective interest sub-dimension and .88 for cognitive interest sub-dimension. As the scale score increases, the interest increases.
Attitude Scale Towards Learning | Evaluated at the end of 6 weeks
  Attitude Scale Towards Learning: The scale developed by Çetin et al. was developed to determine students' attitudes. As a result of all validity and reliability analyzes, there are 34 items in total. Of these scale items, 25 are positive and 9 are negative. The five-point Likert scale is "Totally Agree", "Strongly Agree", "Partly Agree", "Disagree", "Strongly Disagree". The highest attitude score that can be obtained from the scale is 170 and the lowest attitude score is 34. As the attitude score increases, the positive attitude increases. The Cronbach Alpha internal consistency coefficient for the scale was found to be 0.94 for the overall scale.
Class participation | Evaluated at the end of 6 weeks.
  Class participation:
  A weekly signature chart was taken from the students and the number of absenteeism in the last week was calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Metin YILDIZ, Asst.Prof.Dr., Principal Investigator — Sakarya University
Locations (1):
- Sakarya University, Sakarya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Keller, J.M. (2010). Motivational design for learning and performance: The ARCS Model approach. New York, NY: Springer.
- [Background] Dinçer, S., & Doğanay, A. (2016). Öğretim materyali'ne ilişkin motivasyon ölçeği (ÖMMÖ) Türkçe uyarlama çalışması. İlköğretim Online, 15(4).
- [Background] Mazer, J., P. (2013). Validity of the Student Interest and Engagement Scales: Associations with student learning outcomes. Communication Studies, 64, 125-140.
- [Background] Akın, A., Uğur, E., &; Akın, Ü. (2015). Derse İlgi Ölçeğinin Türkçe Formu: Geçerlik ve güvenirlik çalışması. K. U. Kastamonu Eğitim Dergisi 23 (4), 1467-1476.
- [Background] ÇETİN, Ş., & ÇETİN, F. (2019). Öğrenmeye yönelik tutum ölçeği (ÖYTÖ) geliştirme çalışması. Türk Eğitim Bilimleri Dergisi, 17(1), 140-157.